CLINICAL TRIAL: NCT01346488
Title: The Documentation of the Effects on Quality of Life (QOL) and Working Productivity and Activity Impairment (WPAI) in Patients With Rheumatoid Arthritis (RA) Under HUMIRA® (Adalimumab) in Routine Clinical Practice
Brief Title: Special Investigation in Patients With Rheumatoid Arthritis (Working Productivity Activity Impairment)
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-772
Record Dates: First submitted 2011-04-29; First posted 2011-05-03 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Adalimumab: Participants with RA treated with adalimumab who are either engaged in paid work for more than 35 hours per week (paid workers) or those who are either engaged in paid work for less than 35 hours per week or who perform basic activities of daily life other than paid work (home workers).

SUMMARY:
This is a single-arm, multi-center, prospective cohort study (post-marketing observational study). The observation period for each participant is 48 weeks.

This study is designed to provide additional data on treatment effects of adalimumab during 48 weeks of treatment in patients with RA under conditions of routine rheumatology care. Course of work productivity and work ability, the course of health-related quality of life, and changes in functionality during 48 weeks treatment with adalimumab are to be documented.

DETAILED DESCRIPTION:
This study was designed as a non-interventional observational study. Adalimumab was prescribed in the usual manner in accordance with the terms of the local market authorization with regards to dose, population and indication as well as local guidelines.

ELIGIBILITY:
Inclusion Criteria:

RA patients treated with adalimumab who satisfied the following conditions:

1. Paid worker (PW) RA patients who are engaged in paid work for more than 35 hours per week
2. Home worker (HW)

   * Category 1 unpaid workers; RA patients who are engaged in paid work for less than 35 hours per week
   * Category 2 unpaid workers; RA patients who perform basic activities of daily life (household duties, shopping, child caring, exercise, study, etc.) other than PW

Exclusion Criteria:

1. RA patients showing lowered basic activities of daily life, such as hospitalization and being bedridden
2. RA patients with a history of previous treatment with adalimumab

Ages: 15 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Single-arm, Multi-center, Prospective Cohort
Sampling Method: Non-Probability Sample
Enrollment: 2088 (Actual)
Dates: Start 2011-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarina Kurimoto, MD, Study Director — AbbVie

REFERENCES:
- [Result] A Large-Scale Prospective Single Cohort Observational Study of Work Productivity and Activity Impairment In Japanese Patients With Rheumatoid Arthritis Receiving Adalimumab: The Final Analysis of 48-Week Data From the ANOUVEAU Study. EULAR2016 (9 June 2016), poster no. THU0159.
- [Result] Tanaka Y, Yamazaki K, Nakajima R, Komatsu S, Igarashi A, Tango T, Takeuchi T. Economic impact of adalimumab treatment in Japanese patients with rheumatoid arthritis from the adalimumab non-interventional trial for up-verified effects and utility (ANOUVEAU) study. Mod Rheumatol. 2018 Jan;28(1):39-47. doi: 10.1080/14397595.2017.1341459. Epub 2017 Jul 13. PMID 28704126
- [Derived] Takeuchi T, Nakajima R, Komatsu S, Yamazaki K, Nakamura T, Agata N, Igarashi A, Tango T, Tanaka Y. Impact of Adalimumab on Work Productivity and Activity Impairment in Japanese Patients with Rheumatoid Arthritis: Large-Scale, Prospective, Single-Cohort ANOUVEAU Study. Adv Ther. 2017 Mar;34(3):686-702. doi: 10.1007/s12325-017-0477-z. Epub 2017 Jan 31. PMID 28144917
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data sources in this study are from medical charts. Investigators in this study transcribed a participant's data from medical charts to a case report form (CRF) developed by AbbVie.
Pre-assignment Details: A total of 2088 participants filled out registration forms. A total of 1973 participant CRFs were retrieved for use in the study, and 1968 of these were included in the analysis.
Groups:
- Participants Receiving Adalimumab: Participants with rheumatoid arthritis (RA) treated with adalimumab who are either engaged in paid work for more than 35 hours per week (paid workers) or those who are either engaged in paid work for less than 35 hours per week or who perform basic activities of daily life other than paid work (home workers).
Period: Overall Study
Arm/Group | Participants Receiving Adalimumab
Started | 1968
Completed | 1262
Not Completed | 706

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (all evaluable participant CRFs)
Groups:
- Participants Receiving Adalimumab: Participants with RA treated with adalimumab who are either engaged in paid work for more than 35 hours per week (paid workers) or those who are either engaged in paid work for less than 35 hours per week or who perform basic activities of daily life other than paid work (home workers).
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 1968
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1484
  Male | 484

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Work Productivity and Activity Impairment-Rheumatoid Arthritis (WPAI-RA) Questionnaire: Mean Percentage of Work Time Missed (Absenteeism)
Description: Absenteeism, presented as the mean percentage of work time missed due to RA (as reported on the WPAI-RA), and calculated as: 100*number of hours of work missed due to RA / (number of hours of work missed due to RA + number of hours worked). WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. "Change" was calculated as the value at baseline minus the value at each subsequent time point.
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, at discontinuation of adalimumab (ADA) therapy, and at final assessment (up to Week 48)
Population: Participants with evaluable WPAI-RA assessments; number analyzed=participants with an evaluable assessment at given time point.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 782
percentage of work time missed
  Baseline | 7.23 (18.90)
  Change at Week 12: number analyzed (Participants) | 654
  Change at Week 12 | 3.80 (17.61)
  Change at Week 24: number analyzed (Participants) | 547
  Change at Week 24 | 3.73 (16.56)
  Change at Week 36: number analyzed (Participants) | 414
  Change at Week 36 | 3.85 (15.79)
  Change at Week 48: number analyzed (Participants) | 350
  Change at Week 48 | 4.48 (17.91)
  Change at ADA discontinuation: number analyzed (Participants) | 155
  Change at ADA discontinuation | 1.25 (14.46)
  Change at final assessment | 4.23 (17.77)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Week 12; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Week 24; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Week 36; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Week 48; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 5: Comparison: Participants Receiving Adalimumab; at discontinuation of ADA therapy; Test type: Superiority or Other; p = 1.0000, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 6: Comparison: Participants Receiving Adalimumab; at final assessment; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity

2. Primary Outcome: Change From Baseline in WPAI Questionnaire: Mean Percentage of Impairment While Working Due to RA (Presenteeism)
Description: Presenteeism (the extent to which RA decreased productivity) is presented as the mean percentage of impairment while working due to RA, and calculated as: 100*scale value of question 5 on the WPAI (between 0 and 10) / 10. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. "Change" was calculated as the value at baseline minus the value at each subsequent time point.
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, at discontinuation of ADA therapy, and at final assessment (up to Week 48)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 858
percentage of impairment while working
  Baseline | 39.60 (28.53)
  Change at Week 12: number analyzed (Participants) | 731
  Change at Week 12 | 17.18 (26.45)
  Change at Week 24: number analyzed (Participants) | 610
  Change at Week 24 | 20.20 (27.54)
  Change at Week 36: number analyzed (Participants) | 477
  Change at Week 36 | 22.18 (28.37)
  Change at Week 48: number analyzed (Participants) | 397
  Change at Week 48 | 23.32 (27.27)
  Change at ADA discontinuation: number analyzed (Participants) | 174
  Change at ADA discontinuation | 7.64 (29.87)
  Change at final assessment | 19.30 (29.02)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Week 12; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Week 24; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Week 36; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Week 48; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 5: Comparison: Participants Receiving Adalimumab; at discontinuation of ADA therapy; Test type: Superiority or Other; p = 0.0054, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 6: Comparison: Participants Receiving Adalimumab; at final assessment; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity

3. Primary Outcome: Change From Baseline in WPAI Questionnaire: Mean Percentage of Overall Work Productivity Impairment (OWPI) Due to RA
Description: The mean percentage of OWPI due to RA (based on the WPAI questionnaire) is presented, calculated as: Absenteeism (%) + extent to which RA decreased productivity (%)* [number of hours worked / (number of hours of work missed due to RA + number of hours worked)]. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. "Change" was calculated as the value at baseline minus the value at each subsequent time point.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of OWPI
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 771
percentage of OWPI
  Baseline | 41.06 (29.58)
  Change at Week 12: number analyzed (Participants) | 640
  Change at Week 12 | 17.08 (27.60)
  Change at Week 24: number analyzed (Participants) | 536
  Change at Week 24 | 20.83 (28.83)
  Change at Week 36: number analyzed (Participants) | 410
  Change at Week 36 | 22.31 (29.42)
  Change at Week 48: number analyzed (Participants) | 341
  Change at Week 48 | 24.40 (28.37)
  Change at ADA discontinuation: number analyzed (Participants) | 151
  Change at ADA discontinuation | 6.30 (29.60)
  Change at final assessment | 19.77 (29.99)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Week 12; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Week 24; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Week 36; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Week 48; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 5: Comparison: Participants Receiving Adalimumab; at discontinuation of ADA therapy; Test type: Superiority or Other; p = 0.0592, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 6: Comparison: Participants Receiving Adalimumab; at final assessment; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity

4. Primary Outcome: Change From Baseline in WPAI Questionnaire: Mean Percentage of Activity Impairment Due to RA
Description: Activity impairment due to RA (the extent to which RA affected the ability to perform usual daily activities) is presented as the mean percentage of activity impairment, calculated as 100*scale value of WPAI question 6 (between 0 and 10) / 10. WPAI is a questionnaire used to evaluate lost productivity; scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. "Change" was calculated as the value at baseline minus the value at each subsequent time point.
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, at discontinuation of ADA therapy, and final assessment (up to Week 48)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 1546
percentage of activity impairment
  Baseline | 48.42 (28.11)
  Change at Week 12: number analyzed (Participants) | 1339
  Change at Week 12 | 19.42 (25.86)
  Change at Week 24: number analyzed (Participants) | 1113
  Change at Week 24 | 23.30 (28.07)
  Change at Week 36: number analyzed (Participants) | 846
  Change at Week 36 | 25.53 (27.91)
  Change at Week 48: number analyzed (Participants) | 733
  Change at Week 48 | 26.33 (28.17)
  Change at ADA discontinuation: number analyzed (Participants) | 338
  Change at ADA discontinuation | 11.42 (29.83)
  Change at final assessment | 22.36 (29.44)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Week 12; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Week 24; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Week 36; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Week 48; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 5: Comparison: Participants Receiving Adalimumab; at discontinuation of ADA therapy; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 6: Comparison: Participants Receiving Adalimumab; at final assessment; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity

5. Primary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score
Description: The HAQ-DI is a patient-reported questionnaire specific for RA. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 (no disability) to 3 (very severe, high-dependency disability). A negative change from Baseline in the score indicates improvement.
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, at discontinuation of ADA therapy, and final assessment (up to Week 48)
Population: Participants with evaluable HAQ-DI assessments; number analyzed=participants with an evaluable assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 1595
units on a scale
  Baseline | 0.93 (0.75)
  Change at Week 12: number analyzed (Participants) | 1413
  Change at Week 12 | 0.34 (0.51)
  Change at Week 24: number analyzed (Participants) | 1182
  Change at Week 24 | 0.41 (0.55)
  Change at Week 36: number analyzed (Participants) | 912
  Change at Week 36 | 0.42 (0.55)
  Change at Week 48: number analyzed (Participants) | 779
  Change at Week 48 | 0.44 (0.54)
  Change at ADA discontinuation: number analyzed (Participants) | 364
  Change at ADA discontinuation | 0.21 (0.58)
  Change at final assessment | 0.38 (0.57)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Week 12; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Week 24; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Week 36; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Week 48; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 5: Comparison: Participants Receiving Adalimumab; at discontinuation of ADA therapy; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 6: Comparison: Participants Receiving Adalimumab; at final assessment; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity

6. Primary Outcome: Number of Participants Per Category of the HAQ-DI
Description: The HAQ-DI is a patient-reported questionnaire specific for RA. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 (no disability) to 3 (very severe, high-dependency disability). Categories were defined as: high (> 1.5), moderate (≤ 1.5 to > 1.0), low (≤ 1.0 to > 0.5), remission (≤ 0.5 to > 0), 0 (0).
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, at discontinuation of ADA therapy, and final assessment (up to Week 48)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 1595
Participants
  Baseline: High | 326
  Baseline: Moderate | 253
  Baseline: Low | 416
  Baseline: Remission | 411
  Baseline: 0 | 189
  Week 12: number analyzed (Participants) | 1413
  Week 12: High | 135
  Week 12: Moderate | 164
  Week 12: Low | 286
  Week 12: Remission | 417
  Week 12: 0 | 411
  Week 24: number analyzed (Participants) | 1182
  Week 24: High | 94
  Week 24: Moderate | 106
  Week 24: Low | 195
  Week 24: Remission | 354
  Week 24: 0 | 433
  Week 36: number analyzed (Participants) | 912
  Week 36: High | 62
  Week 36: Moderate | 68
  Week 36: Low | 129
  Week 36: Remission | 284
  Week 36: 0 | 369
  Week 48: number analyzed (Participants) | 779
  Week 48: High | 44
  Week 48: Moderate | 57
  Week 48: Low | 115
  Week 48: Remission | 223
  Week 48: 0 | 340
  At discontinuation of ADA therapy: number analyzed (Participants) | 364
  At discontinuation of ADA therapy: High | 69
  At discontinuation of ADA therapy: Moderate | 59
  At discontinuation of ADA therapy: Low | 88
  At discontinuation of ADA therapy: Remission | 78
  At discontinuation of ADA therapy: 0 | 70
  At final assessment: High | 158
  At final assessment: Moderate | 153
  At final assessment: Low | 280
  At final assessment: Remission | 421
  At final assessment: 0 | 583
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Week 12 (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Week 24 (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Week 36 (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Week 48 (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 5: Comparison: Participants Receiving Adalimumab; at discontinuation of ADA therapy (Remission); Test type: Superiority or Other; p = 0.0005, McNemar — P-value adjusted for multiplicity
Statistical Analysis 6: Comparison: Participants Receiving Adalimumab; at final assessment (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity

7. Secondary Outcome: Change From Baseline in Disease Activity Score 28-4 C-Reactive Protein (DAS 28-4 CRP)
Description: DAS28-4 CRP was calculated using the number of tender and swollen joints (out of 28 counted), CRP level, and the participant's global assessment of disease activity via a visual analog scale (VAS). The calculated range of DAS28-4 is 0 (no disease activity) to 10 (maximal disease activity). A decrease from Baseline in score indicates improvement of disease activity.
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, at discontinuation of ADA therapy, and final assessment (up to Week 48)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 1689
units on a scale
  Baseline | 4.20 (1.26)
  Change at Week 12: number analyzed (Participants) | 1500
  Change at Week 12 | 1.55 (1.23)
  Change at Week 24: number analyzed (Participants) | 1282
  Change at Week 24 | 1.81 (1.25)
  Change at Week 36: number analyzed (Participants) | 1077
  Change at Week 36 | 1.91 (1.30)
  Change at Week 48: number analyzed (Participants) | 920
  Change at Week 48 | 2.01 (1.26)
  Change at ADA discontinuation: number analyzed (Participants) | 472
  Change at ADA discontinuation | 0.91 (1.39)
  Change at final assessment | 1.71 (1.39)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Week 12; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Week 24; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Week 36; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Week 48; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 5: Comparison: Participants Receiving Adalimumab; at discontinuation of ADA therapy; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 6: Comparison: Participants Receiving Adalimumab; at final assessment; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity

8. Secondary Outcome: Number of Participants Per Category of the DAS28-4 CRP
Description: DAS28-4 CRP was calculated using the number of tender and swollen joints (out of 28 counted), CRP level, and the participant's global assessment of disease activity via a VAS. The calculated range of DAS28-4 is 0 (no disease activity) to 10 (maximal disease activity). Categories were defined as: high (> 5.1), moderate (≤ 5.1 to > 3.2), low (≤ 3.2 to ≥ 2.6), remission (< 2.6).
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, at discontinuation of ADA therapy, and final assessment (up to Week 48)
Population: Participants with evaluable DAS28-4 CRP assessments; number analyzed=participants with an evaluable assessment at given time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 1689
Participants
  Baseline: High | 402
  Baseline: Moderate | 911
  Baseline: Low | 199
  Baseline: Remission | 177
  Week 12: number analyzed (Participants) | 1500
  Week 12: High | 65
  Week 12: Moderate | 356
  Week 12: Low | 233
  Week 12: Remission | 846
  Week 24: number analyzed (Participants) | 1282
  Week 24: High | 23
  Week 24: Moderate | 203
  Week 24: Low | 203
  Week 24: Remission | 853
  Week 36: number analyzed (Participants) | 1077
  Week 36: High | 11
  Week 36: Moderate | 152
  Week 36: Low | 139
  Week 36: Remission | 775
  Week 48: number analyzed (Participants) | 920
  Week 48: High | 4
  Week 48: Moderate | 96
  Week 48: Low | 117
  Week 48: Remission | 703
  At ADA discontinuation: number analyzed (Participants) | 472
  At ADA discontinuation: High | 76
  At ADA discontinuation: Moderate | 181
  At ADA discontinuation: Low | 61
  At ADA discontinuation: Remission | 154
  At final assessment: High | 91
  At final assessment: Moderate | 319
  At final assessment: Low | 215
  At final assessment: Remission | 1064
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Week 12 (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Week 24 (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Week 36 (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Week 48 (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 5: Comparison: Participants Receiving Adalimumab; at discontinuation of ADA therapy (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 6: Comparison: Participants Receiving Adalimumab; at final assessment (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity

9. Secondary Outcome: Change From Baseline in DAS28-4 Erythrocyte Sedimentation Rate (ESR)
Description: DAS28-4 ESR, a combined index that measures activity of RA, was calculated based on the number of tender and swollen joints (out of 28 counted), general health evaluated by a VAS, and ESR. DAS28-4 ESR scores ranged from 0 (no disease activity) to 10 (maximal disease activity). A decrease from Baseline in scores indicates improvement of disease activity.
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, at discontinuation of ADA therapy, and final assessment (up to Week 48)
Population: Participants with evaluable DAS28-4 ESR assessments; number analyzed=participants with an evaluable assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 1403
units on a scale
  Baseline | 4.76 (1.35)
  Change at Week 12: number analyzed (Participants) | 1241
  Change at Week 12 | 1.61 (1.28)
  Change at Week 24: number analyzed (Participants) | 1058
  Change at Week 24 | 1.91 (1.34)
  Change at Week 36: number analyzed (Participants) | 889
  Change at Week 36 | 2.01 (1.35)
  Change at Week 48: number analyzed (Participants) | 767
  Change at Week 48 | 2.08 (1.33)
  Change at ADA discontinuation: number analyzed (Participants) | 381
  Change at ADA discontinuation | 0.97 (1.43)
  Change at final assessment | 1.80 (1.45)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Week 12; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Week 24; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Week 36; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Week 48; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 5: Comparison: Participants Receiving Adalimumab; at discontinuation of ADA therapy; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 6: Comparison: Participants Receiving Adalimumab; at final assessment; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity

10. Secondary Outcome: Number of Participants Per Category of the DAS28-4 ESR
Description: DAS28-4 ESR, a combined index that measures activity of RA, was calculated based on the number of tender and swollen joints (out of 28 counted), general health evaluated by a VAS, and ESR. DAS28-4 ESR scores ranged from 0 (no disease activity) to 10 (maximal disease activity). Categories were defined as: high (> 5.1), moderate (≤ 5.1 to > 3.2), low (≤ 3.2 to ≥ 2.6), remission (< 2.6).
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, at discontinuation of ADA therapy, and final assessment (up to Week 48)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 1403
Participants
  Baseline: High | 564
  Baseline: Moderate | 662
  Baseline: Low | 101
  Baseline: Remission | 76
  Week 12: number analyzed (Participants) | 1241
  Week 12: High | 113
  Week 12: Moderate | 437
  Week 12: Low | 223
  Week 12: Remission | 468
  Week 24: number analyzed (Participants) | 1058
  Week 24: High | 47
  Week 24: Moderate | 311
  Week 24: Low | 183
  Week 24: Remission | 517
  Week 36: number analyzed (Participants) | 889
  Week 36: High | 33
  Week 36: Moderate | 226
  Week 36: Low | 163
  Week 36: Remission | 467
  Week 48: number analyzed (Participants) | 767
  Week 48: High | 16
  Week 48: Moderate | 169
  Week 48: Low | 135
  Week 48: Remission | 447
  At ADA discontinuation: number analyzed (Participants) | 381
  At ADA discontinuation: High | 96
  At ADA discontinuation: Moderate | 165
  At ADA discontinuation: Low | 39
  At ADA discontinuation: Remission | 81
  At final assessment: High | 124
  At final assessment: Moderate | 398
  At final assessment: Low | 227
  At final assessment: Remission | 654
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Week 12 (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Week 24 (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Week 36 (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Week 48 (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 5: Comparison: Participants Receiving Adalimumab; at discontinuation of ADA therapy (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 6: Comparison: Participants Receiving Adalimumab; at final assessment (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity

11. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI)
Description: The CDAI is a validated measure of RA disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, global health assessed by the participant on a VAS from 0 to 10 (cm), and global health assessed by an investigator on a visual analogue scale from 0 to 10 (cm) were included in the CDAI score. Scores on the CDAI range from 0 (lowest disease activity) to 76 (highest disease activity). "Change" was calculated as the value at baseline minus the value at each subsequent time point.
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, at discontinuation of ADA therapy, and final assessment (up to Week 48)
Population: Participants with evaluable CDAI assessments; number analyzed=participants with an evaluable assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 1696
units on a scale
  Baseline | 21.44 (12.24)
  Change at Week 12: number analyzed (Participants) | 1515
  Change at Week 12 | 11.98 (11.06)
  Change at Week 24: number analyzed (Participants) | 1296
  Change at Week 24 | 13.93 (11.12)
  Change at Week 36: number analyzed (Participants) | 1079
  Change at Week 36 | 14.26 (11.56)
  Change at Week 48: number analyzed (Participants) | 916
  Change at Week 48 | 14.63 (11.19)
  Change at discontinuation of ADA therapy: number analyzed (Participants) | 485
  Change at discontinuation of ADA therapy | 8.00 (12.14)
  Change at final assessment | 12.94 (12.11)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Week 12; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Week 24; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Week 36; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Week 48; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 5: Comparison: Participants Receiving Adalimumab; at discontinuation of ADA therapy; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 6: Comparison: Participants Receiving Adalimumab; at final assessment; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity

12. Secondary Outcome: Number of Participants Per Category of the CDAI
Description: The CDAI is a validated measure of RA disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, global health assessed by the participant on a VAS from 0 to 10 (cm), and global health assessed by an investigator on a visual analogue scale from 0 to 10 (cm) were included in the CDAI score. Scores on the CDAI range from 0 (lowest disease activity) to 76 (highest disease activity). Categories were defined as: high (> 22.1), moderate (≤ 22.0 to > 10.0), low (≤ 10.0 to < 2.8), and remission (≤ 2.8).
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, at discontinuation of ADA therapy, and final assessment (up to Week 48)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 1696
Participants
  Baseline: High | 677
  Baseline: Moderate | 749
  Baseline: Low | 249
  Baseline: Remission | 21
  Week 12: number analyzed (Participants) | 1515
  Week 12: High | 128
  Week 12: Moderate | 374
  Week 12: Low | 676
  Week 12: Remission | 337
  Week 24: number analyzed (Participants) | 1296
  Week 24: High | 51
  Week 24: Moderate | 245
  Week 24: Low | 595
  Week 24: Remission | 405
  Week 36: number analyzed (Participants) | 1079
  Week 36: High | 34
  Week 36: Moderate | 183
  Week 36: Low | 459
  Week 36: Remission | 403
  Week 48: number analyzed (Participants) | 916
  Week 48: High | 19
  Week 48: Moderate | 113
  Week 48: Low | 384
  Week 48: Remission | 400
  At ADA discontinuation: number analyzed (Participants) | 485
  At ADA discontinuation: High | 114
  At ADA discontinuation: Moderate | 171
  At ADA discontinuation: Low | 138
  At ADA discontinuation: Remission | 62
  At final assessment: High | 149
  At final assessment: Moderate | 338
  At final assessment: Low | 639
  At final assessment: Remission | 570
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Week 12 (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Week 24 (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Week 36 (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Week 48 (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 5: Comparison: Participants Receiving Adalimumab; at discontinuation of ADA therapy (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity
Statistical Analysis 6: Comparison: Participants Receiving Adalimumab; at final assessment (Remission); Test type: Superiority or Other; p < 0.0001, McNemar — P-value adjusted for multiplicity

13. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions Questionnaire (EQ-5D) Summary Index Score
Description: The EQ-5D is a participant answered questionnaire scoring 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. EQ-5D health states, defined by the EQ-5D descriptive system, are converted into a single summary index by applying a formula that essentially attaches values (also called QOL weights or QOL utilities) to each of the levels in each dimension. EQ-5D Summary Index values range from -0.594 to 1 (with higher scores indicating better health state). "Change" was calculated as the value at baseline minus the value at each subsequent time point.
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, at discontinuation of ADA therapy, and final assessment (up to Week 48)
Population: Participants with evaluable EQ-5D assessments; number analyzed=participants with an evaluable assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 1566
units on a scale
  Baseline | 0.6295 (0.1545)
  Change at Week 12: number analyzed (Participants) | 1370
  Change at Week 12 | -0.1112 (0.1651)
  Change at Week 24: number analyzed (Participants) | 1151
  Change at Week 24 | -0.1380 (0.1805)
  Change at Week 36: number analyzed (Participants) | 881
  Change at Week 36 | -0.1574 (0.1836)
  Change at Week 48: number analyzed (Participants) | 765
  Change at Week 48 | -0.1541 (0.2020)
  Change at discontinuation of ADA therapy: number analyzed (Participants) | 349
  Change at discontinuation of ADA therapy | -0.0597 (0.1577)
  Change at final assessment | -0.1356 (0.1908)
Statistical Analysis 1: Comparison: Participants Receiving Adalimumab; Week 12; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 2: Comparison: Participants Receiving Adalimumab; Week 24; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 3: Comparison: Participants Receiving Adalimumab; Week 36; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 4: Comparison: Participants Receiving Adalimumab; Week 48; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 5: Comparison: Participants Receiving Adalimumab; at discontinuation of ADA therapy; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity
Statistical Analysis 6: Comparison: Participants Receiving Adalimumab; at final assessment; Test type: Superiority or Other; p < 0.0001, Paired t-test — P-value adjusted for multiplicity

14. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), and Deaths
Description: AEs, which were defined as any untoward medical occurrence observed in participants who received adalimumab in this study, were summarized.
Time Frame: up to Week 52
Population: Safety Analysis Set (all evaluable participants with validated CRFs)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 1968
Participants
  AEs | 475
  SAEs | 103
  Deaths | 5

15. Secondary Outcome: Number of Participants With Adverse Drug Reactions
Description: Adverse drug reactions were defined as AEs of which a causal relationship with adalimumab could not be ruled out.
Time Frame: up to Week 52
Population: Safety Analysis Set (all evaluable participants with validated CRFs)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Adalimumab
Number analyzed (Participants) | 1968
Participants | 451

ADVERSE EVENTS:
Time Frame: up to Week 52
Description: Safety of adalimumab therapy was assessed using data obtained from the day of the first administration to 52 weeks after the initiation of adalimumab therapy. (Although adalimumab was administered for 48 weeks in this study, data during the 4 weeks after the end of Week 48 were also included into the analysis for participants for whom data after the treatment was described in their CRFs).
Arm/Group | Participants Receiving Adalimumab
Serious Adverse Events (participants affected / at risk) | 103/1968
Other Adverse Events (participants affected / at risk) | 202/1968
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Receiving Adalimumab (N=1968)
Appendicitis (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 2
Meningitis salmonella (Infections and infestations) | 1
Meningitis viral (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 9
Pneumonia mycoplasmal (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Muscle abscess (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Bacterial sepsis (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 2
Bursitis infective (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 5
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemangioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Meningioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Follicle centre lymphoma, follicular grade I, II, III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancytopenia (Blood and lymphatic system disorders) | 2
Completed suicide (Psychiatric disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 3
Subarachnoid haemorrhage (Nervous system disorders) | 1
Cataract (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Polypoidal choroidal vasculopathy (Eye disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Aortic aneurysm rupture (Vascular disorders) | 1
Rheumatoid vasculitis (Vascular disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 8
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
Death (General disorders) | 1
Pyrexia (General disorders) | 3
White blood cell count decreased (Investigations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 3
Femur fracture (Injury, poisoning and procedural complications) | 5
Humerus fracture (Injury, poisoning and procedural complications) | 1
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Receiving Adalimumab (N=1968)
Bronchitis (Infections and infestations) | 27
Nasopharyngitis (Infections and infestations) | 32
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 28
Hepatic function abnormal (Hepatobiliary disorders) | 59
Rash (Skin and subcutaneous tissue disorders) | 34
Injection site erythema (General disorders) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.